CLINICAL TRIAL: NCT05393024
Title: Observational Study in Patient With Multiple Myeloma Relapse/Refractory Treated With Belantamab Mafotidine on Monotherapy Previously Exposed to at Least One Proteasome Inhibitor, Immunomodulatory Agent, and Anti-CD38 Antibody.
Brief Title: Patient With MMRR Treated With Belantamab Mafotidine on Monotherapy
Status: Completed | Type: Observational
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: REAL-BELAMAF-ITALY
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Mulitple Myeloma; Belantamab Mafoditin; EAP
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Belantamab Mafoditin: MMRR patients included in Named Patient Program and Expanded Access Program
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — MMRR patients included in Named Patient Program e Expanded Access Program

SUMMARY:
This is a retrospective/prospective observational study evaluating the efficacy and safety of Belantamab Mafotidin as a single agent in patients with Multiple Myeloma Relapse/Refractory (MMRR) treated in clinical pratice under compassionate use

DETAILED DESCRIPTION:
Multiple myeloma (MM) is an incurable disease that accounts for 1% of all cancers and 10% of all haematological malignancies, most patients with MM develop resistance to existing therapies at the time of disease recurrence.

Belantamab mafodotin is a new humanized antibody-drug conjugate (IgG1) that is under development for the treatment of MM and has demonstrated a manageable safety profile and positive clinical activity in patients with relapsed or refractory multiple myeloma (MMRR) heavily pretreated.

The objective of this retro-prospective observational study is: to evaluate clinical efficacy as the percentage of patients who have achieved a clinical benefit (minimum or best response), ORR, DoR, PFS, OS; evaluate the safety profile of patients treated with Belantamab Mafodotin as monotherapy in clinical practice.

All patients included in this analysis were treated or are still receiving Belantamab Mafodotin monotherapy under the compassionate use programs (nominal program-NPP and the extended access program-EAP).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent may be obtained from the patient or legally authorized representative according to local regulations (patients who have already died may also be included)
2. Histologically or cytologically confirmed diagnosis of MM as defined according to IMWG criteria of 2016 and:

   1. patient has undergone stem cells transplantation or is considered ineligible for transplantation, and
   2. patient has received at least four therapies
   3. patient is refractory to an anti-CD38 antibody (ex., daratumumab) alone or in combination, and to an IMiD (ex., lenalidomide or pomalidomide), and to a proteasome inhibitor (ex. bortezomib, ixazomib or carfilzomib).
3. Male or female equal and/or upper 18 years (at baseline)
4. Performance Status at baseline by ECOG scale 0-2
5. Adequate organ system functions at baseline
6. Female patients: a female patient is elegible if she is not pregnant or breastfeeding and at least one of the following conditions applies:

   * She is/was not a woman of childbearing potential (WOCBP) OR
   * She is/was using an highly effective contrapcetive method during the treatment period and at least 9 months after the last dose and she agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period.
   * Highly sensitive negative serum pregnancy test within 72 hours of therapy (C1D1) and agreed to use effective contraception during the treatment period and for the next 9 months after the last dose of the drug.

   Male patient: male patient were/are elegible if agreed to follow from the first dose until the last dose of treatment to allow clearance of any altered sperm:
   * abstaining from sperm donation PLUS
   * abstaing from heterosexual relationship in accordance with one's preferred and habitual lifestyle (long-term and persistent abstinent) and agreed/accepted to remain abstinent OR
   * agree/agreed to use contraption as described below: agree to use male condom even though they have/had succesfully vasectomy and female partner uses/used an additional highly effective contraceptive method.
7. All toxicities related to previous treatment (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE) were Grade 1 or less at t at the time of treatment initiation within compassionate use programs, except alopecia and neuropathy grade 2.

Exclusion Criteria:

* The patients are/were not elegible for compassionate use programs (NPP, EAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with MMRR previously treated with at least one proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 antibody.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Best response or minimal response | 1 year
  percentage of patients that achieved a clinical benefit

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  percertange of patient with confirmed partial response
Progression Free Survival (PFS) | 1 year
  time from the first Belantamab Mafodotin administration until disease progression
Duration of Response (DoR) | 1 year
  time for first documentated partial or best response until disease progression
Overall Survival | 1 year
  time from starting of treatment until death or other cause

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Petrucci, MD, Principal Investigator — Policlinico Umberto I - Università 'Sapienza'; Massimo Offidani, MD, Principal Investigator — A.O.U. Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi di Ancona
Locations (10):
- Italy (10):
  - AOU Ospedali Riuniti Umberto I, Ancona
  - Policlinico Sant'Orsola Malpighi, Aou Di Bologna, Bologna
  - A.O. Spedali Civili di Brescia, Brescia
  - Ospedale "A. Businco", Cagliari
  - AOU Policlinico Vittorio Emanuele, Catania
  - A.O.U. Arcispedale Sant'Anna, Ferrara
  - Fondazione IRCCS Ca' Grande Ospedale Maggiore Policlinico, Milan
  - A.O.U. Federico II, Napoli
  - La Maddalena S.p.a, Palermo
  - Policlinico Umberto I - Università La Sapienza, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Result] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245